CLINICAL TRIAL: NCT02685332
Title: Phase I Dose Escalation Trial of Single Fraction Adjuvant Stereotactic Body Partial Breast Irradiation (SB-PBI) For Early Stage Breast Cancer
Brief Title: Phase I Dose Escalation of Single Fraction Adjuvant Stereotactic Body Partial Breast Irradiation Early Stage Breast CA
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Asal Rahimi, ASSOC PROFESSOR, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STU 062015-085
Record Dates: First submitted 2016-02-11; First posted 2016-02-18 (Estimated); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Early Stage Breast Cancer
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (1):
- Stereotactic Radiation (Experimental): Single Fraction Stereotactic Radiation. Step No. Fractions Dose per fraction
  -1 1 20 0 (starting) 1 22.5
  1. 1 26.5
  2. 1 30
  Interventions: Radiation: Stereotactic Radiation

INTERVENTIONS:
Radiation: Stereotactic Radiation — Stereotactic Body Partial Breast irradiation Step No. Fractions Dose per fraction
  -1 1 20 0 (starting) 1 22.5
  1. 1 26.5
  2. 1 30
  Other Names: SB-PBI

SUMMARY:
Radiation, Stereotactic Body Radiation Therapy.

DETAILED DESCRIPTION:
In this protocol, we plan to use the uniqueness of the Cyberknife system to deliver an adjuvant single fraction radiation dose. We anticipate that this radiation deliver system will reduce toxicity and improve cosmesis. Extrapolating from an intra-operative body of work, this Phase I study will attempt to achieve a non-invasive low toxicity profile and maintain good to excellent cosmesis. In this effort, the Cyberknife system will be used to achieve high conformality and dose gradient.

ELIGIBILITY:
Inclusion Criteria:

* Ductal carcinoma in situ (DCIS) or invasive epithelial (ductal, medullary, papillary, mucinous (colloid), or tubular histologies
* Willing and able to provide consent
* Age >=18 years.
* Performance status Eastern Cooperative Oncology Group (ECOG) 0-2
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Appropriate staging studies identifying as American Joint Committee on Cancer (AJCC) stage 0, I, or II breast cancer. If stage II, the tumor size must be 3 cm or less.
* Surgical treatment of the breast with lumpectomy Clinical Target Volume (CTV) margin up to 5 cm in maximum dimension with histologically confirmed margins free of tumor (negative margins defined as no tumor on ink in all directions). Re-excision of surgical margins is permitted.
* Gross disease within the breast must be unifocal. (Patients with microscopic multifocality are eligible as long as the total extent of tumor, gross and microscopic, occupies a volume with greatest dimension 3 cm or less)
* Patients with invasive disease are required to have axillary staging including: sentinel node biopsy alone if sentinel node is negative, sentinel node biopsy followed by axillary dissection with a minimum of 6 axillary nodes sampled if sentinel node is positive, or axillary dissection alone (with a minimum of 6 axillary nodes). Patients with DCIS are not required to have axillary staging.
* Patients with a history of non-breast invasive malignancies are eligible if they have been disease-free for 1 or more years prior to entry into the study

Exclusion Criteria:

* T2 (>3.0 cm), T3, stage III, or stage IV breast cancer
* More than 3 histologically positive axillary lymph nodes or axillary lymph nodes with microscopic or macroscopic extracapsular extension.
* Positive non-axillary sentinel nodes or evidence of suspicious supraclavicular, infraclavicular, or internal mammary nodes by imaging or physical exam, unless biopsied and found to be negative for tumor.
* Evidence by physical examination or mammography of other suspicious masses, densities, or microcalcifications in either breast, unless biopsied and found to be benign.
* Non epithelial breast malignancies such as sarcoma or lymphoma.
* Multicentric gross breast carcinoma (either DCIS or invasive cancer) or microscopic breast carcinoma occupying a volume with maximum dimensions of more than 3 centimeters.
* Synchronous bilateral invasive or non-invasive breast cancer.
* Paget's disease of the nipple.
* Previous breast radiation on ipsilateral side or thoracic radiation on the ipsilateral side.
* Treatment plan that includes regional nodal irradiation.
* Any prior treatment with radiation therapy or chemotherapy for the currently diagnosed breast cancer prior to registration. Endocrine therapy may be given but not within 28 days prior to study entry and must be stopped if the patient will be receiving chemotherapy until completion of chemotherapy. Patients must discontinue any hormonal agents such as raloxifene, tamoxifen, or other selective estrogen receptor modulators prior to registration.
* Patients with collagen vascular disease, specifically dermatomyositis with a Creatine phosphokinase (CPK) level above normal or active skin rash, systemic lupus erythematosis, or scleroderma.
* Pregnancy or lactation at the time of registration. For women of childbearing age, they must agree to use effective contraceptive methods such as condom/diaphragm and spermicidal foam, intrauterine device, or prescription birth control pills.
* Patients with severe co-extensive comorbidities or significant psychiatric illness.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-03-31 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
maximum tolerated dose | 3 years
  maximum tolerated radiation dose

SECONDARY OUTCOMES:
dose-limiting toxicity | 90 days
  dose-limiting toxicity for each dose level
cosmesis | follow up at month 3, 6, 12, 24, 36, 48, and 60
  as evaluated by an independent panel judging from serial photography

OTHER OUTCOMES:
breast recurrence rate | 5 years
distant disease-free interval | 5 years
  the time from registration to first diagnosis of distant disease
recurrence free survival | 5 years
  time from registration to first diagnosis of a local, regional, or distant recurrence
overall survival | 5 years
  time from registration to death due to any cause
treatment related fibrosis | follow up at month 6, 12, 18, and 24
  Strain elastography, an imaging modality, which will be utilized to determine different degrees of treatment related fibrosis.

CONTACTS AND LOCATIONS:
Overall Officials: Asal Rahimi, MD, Principal Investigator — UTSW Medical Center
Locations (2):
- United States (2):
  - NYU Winthrop Hospital, Mineola, New York
  - The University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No